CLINICAL TRIAL: NCT00704171
Title: Prospective Multi-Center Randomized Post Market Study to Evaluate the PleuraSeal Sealant System as Adjunct to Standard Closure Techniques for Control of Visceral Pleural Air Leaks Following Elective Pulmonary Resection Via Open Thoracotomy
Brief Title: PleuraSeal Post Market Study (Europe)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUN-06-002
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Results first posted 2010-03-15 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Lung Disease; Pulmonary Lobectomy
Keywords: Elective pulmonary resection via open thoracotomy.
MeSH Terms: conditions — Lung Diseases | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PleuraSeal (Experimental): PleuraSeal Lung Sealant System
  Interventions: Device: PleuraSeal Lung Sealant System
- Standard of Care (Active Comparator): Standard tissue closure techniques (control) - sutures or staples only
  Interventions: Procedure: Standard Tissue Closure Techniques; Device: PleuraSeal Lung Sealant System

INTERVENTIONS:
Procedure: Standard Tissue Closure Techniques — Standard Tissue Closure Techniques (sutures and staples only)
  Other Names: Sutures or staples
  Arms: Standard of Care
Device: PleuraSeal Lung Sealant System
  Other Names: PleuraSeal

SUMMARY:
To further characterize the PleuraSeal Sealant System as compared to standard of care (sutures and staples only) in subjects undergoing an elective pulmonary lobectomy and segmentectomy via open thoractomy.

ELIGIBILITY:
Pre-Operative Inclusion Criteria:

* Subjects 18 years of age or older
* Scheduled for an elective pulmonary lobectomy and segmentectomy (limited resection in case of reduced functional operability) in one or more lobes via an open thoracotomy
* Subject or authorized representative has been informed of the nature of the study and has provided written informed consent, approved by the appropriate Ethics Committee of teh respective clinical site

Pre-Operative Exclusion Criteria:

* Documented history of bleeding disorders and/or severely altered renal or hepatic function
* Compromised immune system (e.g., HIV/acquired immunodeficiency syndrome, immunosuppressive therapy)
* Prior ipsilateral thoracotomy
* Subject with Tuberculosis
* Extensive adhesions from previous thoracic trauma or surgery
* Undergoing lung volume reduction surgery, wedge resection, pneumonectomy, sleeve resection or bronchoplasty, blebectomy, bullectomy, pleurodesis, lung transplant, or living lobe transplant donor
* Subject has active systemic or pulmonary infection
* Treated with chronic steroid therapy unless discontinued more than 6 weeks prior to surgery (standard acute perioperative steroids are permitted). For purposes of this protocol, chronic steroid therapy is defined as greater than 4 weeks
* Pregnant (documented by pregnancy test), breast-feeding, or that wish to become pregnant during the course of the study or not willing to use birth control (e.g. IUD; oral, transdermal or parenteral contraceptives; abstinence)
* Documented history of uncontrolled diabetes
* Subject has an estimated life expectancy of less than 6 months
* Currently enrolled in another investigational drug or device trial that has not completed the primary endpoint or that clinically interferes with this study
* Congestive heart failure, cor pulmonale, or other condition that, in the opinion of the investigator, may jeopardize the subject's well-being and/or negatively impact the interpretation of data collected during the clinical study
* Unable to comply with the study requirements or follow-up schedule

Intra-Operative Inclusion Criteria:

* At least one intra-operative air leak identified during lung submersion leak test after the initial closure is completed
* Hemostasis must be confirmed prior to randomization

Intra-Operative Exclusion Criteria:

* Procedure performed via VATS only
* Air leaks originating from bronchioles >1 mm in diameter that cannot be primarily closed or a residual tidal volume loss of >=30%
* Extensive intra-thoracic adhesions present
* Exploratory thoracotomy performed only
* Pneumonectomy, wedge resection, sleeve resection, pleurodesis, bronchoplasty, blebectomy or bullectomy performed
* Incidental finding of any other pre-operative exclusion criteria
* Use of buttressing materials or other non-autologous staple/suture line reinforcement or other surgical sealants when used for pulmonary sealing (i.e., use of hemostatic agents for hemostasis is permitted); however, the sealant should not be applied over intact hemostatic material and all hemostat should be removed prior to sealant application
* Investigator determines that participation in the study may jeopardize the safety or welfare of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Doyle, Study Director — Senior Director, Clinical Affairs at Covidien (formerly Confluent); Paul De Leyn, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (9):
- Covidien, Bedford, Massachusetts, United States
- Austria (2):
  - Universitaetsklinik - Landeskrankenhaus Innsbruck, Innsbruck
  - Otto Wagner Spital, Vienna
- Belgium (2):
  - Hopital Erasme, Brussels
  - University Hospitals Leuven, Leuven
- Netherlands (2):
  - VU-Medisch Centrum, Amsterdam
  - Medical Centre Rotterdam Zuid, Rotterdam
- University Hospital - Zurich, Zurich, Switzerland
- Papworth Hospital, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 28, 2008 and October 21, 2008, a total of 161 subjects were consented and screened for potential study participation at 8 institutions (hospitals). Of these subjects, 121 were randomized.
Pre-assignment Details: Subjects were evaluated for pre-operative and intra-operative eligibility criteria. Randomization occurred intra-operatively.
Period: Overall Study
Arm/Group | PleuraSeal | Standard of Care
Started | 62 | 59
Completed | 61 (One subject withdrew consent prior to study completion. No reason given.) | 59 (All control subjects completed the study.)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PleuraSeal | Standard of Care | Total
Number analyzed (Participants) | 62 | 59 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.1) | 62.8 (10.8) | 62.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 36 | 37 | 73
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 61 | 55 | 116
  African | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Hispanic | 0 | 1 | 1
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Netherlands | 9 | 6 | 15
  Belgium | 14 | 14 | 28
  United Kingdom | 6 | 4 | 10
  Austria | 32 | 30 | 62
  Switzerland | 1 | 5 | 6
Nicotine Use [Number; unit: participants]
  History | 31 | 34 | 65
  Current | 22 | 17 | 39
  Never | 9 | 8 | 17
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.86 (4.73) | 26.35 (4.55) | 26.10 (4.63)
Height [Mean (Standard Deviation); unit: cm] | 169.5 (8.8) | 169.4 (9.6) | 169.4 (9.1)
Weight [Mean (Standard Deviation); unit: kg] | 74.46 (15.35) | 75.57 (13.96) | 75.00 (14.64)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Remaining Air Leak Free From Time of Skin Closure to Hospital Discharge.
Time Frame: 30 days
Measure: Number; unit: Percentage of participants
Arm/Group | PleuraSeal | Standard of Care
Number analyzed (Participants) | 62 | 59
Percentage of participants | 41.9 | 30.5
Statistical Analysis 1: Comparison: PleuraSeal vs Standard of Care; Primary objective was to demonstrate superiority of PleuraSeal as an adjunct compared to standard of care alone. Tissue closure rates for the treatment and control groups were assumed to be 0.40 and 0.15, respectively. To achieve 80 percent power (alpha=0.05, 2-tailed, Fisher's Exact Test) required 112 completed subjects. To account for potential subject withdrawals, an additional 8 subjects were to be enrolled for a total of 120 randomized subjects (approx. 60 per treatment group); Test type: Superiority or Other; p = 0.257, Fisher Exact

2. Secondary Outcome: Percentage of Subjects for Whom Intra-operative Air Leak Sealing Success is Achieved.
Description: Success is defined as no presence of air leak intra-operatively.
Time Frame: Intra-operatively, time of study procedure
Measure: Number; unit: Percentage of participants
Arm/Group | PleuraSeal | Standard of Care
Number analyzed (Participants) | 62 | 59
Percentage of participants | 71 | 23.7
Statistical Analysis 1: Comparison: PleuraSeal vs Standard of Care; Test type: Superiority or Other; p < 0.001, Fisher Exact; two-sided

3. Secondary Outcome: Time From Skin Closure to Last Observable Air Leak.
Time Frame: 30 days
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PleuraSeal | Standard of Care
Number analyzed (Participants) | 62 | 59
hours | 6.0 [0.0 to 30.0] | 30.0 [6.0 to 30.0]
Statistical Analysis 1: Comparison: PleuraSeal vs Standard of Care; Test type: Superiority or Other; p = 0.790, Kaplan-Meier; Kaplan-Meier method was used to obtain estimated median times for each treatment group and the log-rank test was used to compare the two treatments

4. Secondary Outcome: Duration of Chest Drainage
Time Frame: 30 days
Measure: Median (Standard Deviation); unit: hours
Arm/Group | PleuraSeal | Standard of Care
Number analyzed (Participants) | 62 | 59
hours | 93.68 (127.88) | 94.05 (81.05)
Statistical Analysis 1: Comparison: PleuraSeal vs Standard of Care; Test type: Superiority or Other; p = 0.559, 2-sample t-test

5. Secondary Outcome: Duration of Hospitalization
Time Frame: 30 days
Measure: Median (Standard Deviation); unit: hours
Arm/Group | PleuraSeal | Standard of Care
Number analyzed (Participants) | 62 | 59
hours | 312.0 (419.2) | 288.0 (254.1)
Statistical Analysis 1: Comparison: PleuraSeal vs Standard of Care; Test type: Superiority or Other; p = 0.292, 2-sample t-test

6. Primary Outcome: Percentage of Subjects Remaining Air Leak Free From Skin Closure to Discharge
Description: Sub-analysis by pre-randomization grade of air leak. Grade 1= countable air bubbles, Grade 2= stream of bubbles, Grade 3= coalesced bubbles
Time Frame: 30 days
Population: Analysis by grade of air leak.Grade 1= countable air bubbles, Grade 2= Stream of bubbles, Grade 3 = Coalesced bubbles.
Measure: Number; unit: Percentage of participants
Arm/Group | PleuraSeal | Standard of Care
Number analyzed (Participants) | 62 | 59
Percentage of participants
  Grade 1 air leak | 37.5 | 50
  Grade 2/3 air leak | 43.5 | 15.2
Statistical Analysis 1: Comparison: PleuraSeal vs Standard of Care; Test type: Superiority or Other; p = 0.53, Fisher Exact — For subgroup with pre-randomization air leak grade of 1
Statistical Analysis 2: Comparison: PleuraSeal vs Standard of Care; Test type: Superiority or Other; p = .013, Fisher Exact — For subgroup with pre-randomization air leak grade of 2 or 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of randomization until completion of the study, 30 days postoperatively.
Description: Events deemed probable, possible, or definitely related to treatment (PleuraSeal or Control) were to be followed until resolution or 60 days following end of study (whichever comes first).
Arm/Group | PleuraSeal | Standard of Care
Serious Adverse Events (participants affected / at risk) | 16/62 | 11/59
Other Adverse Events (participants affected / at risk) | 2/62 | 4/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PleuraSeal (N=62) | Standard of Care (N=59)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Chronic (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 2 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PleuraSeal (N=62) | Standard of Care (N=59)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator agree to submit the draft of any proposed publication to Sponsor at least 30 dyas prior to submission for publication, presentation, or use, and agrees, at the request of the Sponsor, to withhold any such submission for an additional period, not to exceed 90 days to allow Sponsor to file patent applications. The first publication of the results shall be made in conjunction with the presentation of a joint, multi-center publication.